CLINICAL TRIAL: NCT05265624
Title: A Phase 2 Study of the Value of Pre-symptomatic Genetic Risk Assessment for Age-Related Macular Degeneration
Brief Title: The Moran AMD Genetic Testing Assessment Study
Acronym: MAGENTA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Paul S. Bernstein (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor-Investigator, Paul S. Bernstein, Professor, Ophthalmology/Visual Sciences, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 150093; 1R21EY033579 (NIH)
Record Dates: First submitted 2022-02-08; First posted 2022-03-03 (Actual); Results first posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Age-Related Macular Degeneration; Genetic Testing; Nutritional Biomarkers
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be masked to their AMD risk until their disclosure. Outcomes assessor and investigator will be masked to treatment assignment until completion of study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Genetic Results Disclosure (Experimental): Early disclosure group receives results of genetic testing at Month 1
  Interventions: Behavioral: Early disclosure of genetic testing results
- Late Genetic Results Disclosure (Active Comparator): Late disclosure group receives results of genetic testing at Month 12
  Interventions: Behavioral: Late disclosure of genetic testing results

INTERVENTIONS:
Behavioral: Early disclosure of genetic testing results — Early disclosure group receives results of genetic testing at Month 1
  Arms: Early Genetic Results Disclosure
Behavioral: Late disclosure of genetic testing results — Late disclosure group receives results of genetic testing at Month 12
  Arms: Late Genetic Results Disclosure

SUMMARY:
The goals of this study are:

To assess the impact of genetic testing for Age-related Macular Degeneration (AMD) on lifestyle behaviors as measured by systemic and ocular carotenoid status.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between 18 and 64 years of age.
* They must also be Caucasian as this genetic test is only validated in Caucasians.
* They can have a positive family history of AMD but this is not necessary.

Exclusion Criteria:

* Personal history of AMD
* Non Caucasian
* Employee of the Moran or other eye care practice (likely to have more knowledge about AMD than a layperson)
* Personal history of prior genetic testing for AMD risk
* Anticipated cataract surgery in the upcoming year (can affect Macular Pigment measurement)
* Major psychiatric disorder

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Bernstein, MD, PhD, Principal Investigator — University of Utah Moran Eye Center
Locations (1):
- University of Utah John A. Moran Eye Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Addo EK, Hartnett ME, Bernstein PS. The value of pre-symptomatic genetic risk assessment for age-related macular degeneration: the Moran AMD Genetic Testing Assessment (MAGENTA) study-a study protocol for a randomized controlled trial. Trials. 2023 Jun 19;24(1):414. doi: 10.1186/s13063-023-07436-4. PMID 37337222

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Early Genetic Results Disclosure | Late Genetic Results Disclosure
Started | 60 | 20
Completed | 56 | 20
Not Completed | 4 | 0
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Genetic Results Disclosure | Late Genetic Results Disclosure | Total
Number analyzed (Participants) | 60 | 20 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (10.6) | 51.3 (10.3) | 48.6 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 14 | 63
  Male | 11 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 60 | 20 | 80
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 60 | 20 | 80
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 60 | 20 | 80
Skin carotenoid status at baseline by RS [Mean (Standard Deviation); unit: Reflection Units (RU)] — Reflectance Spectroscopy (RS) is measured by Veggie Meter and is presented in Reflection Units (RU). Possible scores range from 0 (no carotenoids detected) to greater than 500.
  Reflection Units (RU) | 269 (113.5) | 261 (101.1) | 267.5 (110)
Skin carotenoid status at baseline by RRS [Mean (Standard Deviation); unit: Resonance Raman Units (RRU)] — Resonance Raman Spectroscopy (RSS) is presented in Resonance Raman Units (RRU). Possible scores range from 0 (no carotenoids detected) to greater than 100,000.
  Resonance Raman Units (RRU) | 27,865 (9,089.6) | 27,185 (7,470.3) | 27,695.5 (8,672.6)
Macular carotenoid status at baseline [Mean (Standard Deviation); unit: unitless] — Macular Pigment Optical Volume (MPOV) is a unitless measure of the amount of carotenoids present in the macula. Possible scores range from 0 (no carotenoids detected) to greater than 50,000.
  unitless | 10,252 (4,861.3) | 9,945 (4,286.7) | 10,175.5 (4,699.6)
Serum carotenoid status at baseline [Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)] — Serum carotenoid levels are measured in nanograms per milliliter (ng/mL). Possible scores range from 0 (no carotenoids detected) to greater than 1,000.
  nanograms per milliliter (ng/mL) | 623.9 (357.2) | 541.8 (247.3) | 603.3 (333.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Skin Carotenoid Status in Response to Genetic Risk Disclosure as Measured by Reflectance Spectroscopy
Description: Reflectance Spectroscopy (RS) is measured by Reflection Units. Possible scores range from 0 (no carotenoids detected) to greater than 500. Change = (Month 12 Score - Baseline Score).
Time Frame: Baseline and Month 12
Measure: Mean (Standard Error); unit: Reflection units (RU)
Arm/Group | Early Genetic Results Disclosure | Late Genetic Results Disclosure
Number analyzed (Participants) | 56 | 20
Reflection units (RU) | 257.7 (7.4) | 290.9 (12.5)

2. Primary Outcome: Change in Skin Carotenoid Status in Response to Genetic Risk Disclosure as Measured by Resonance Raman Spectroscopy
Description: Resonance Raman Spectroscopy (RSS) is measured in Resonance Raman Units (RRU). Possible scores range from 0 (no carotenoids detected) to greater than 100,000. Change = (Month 12 Score - Baseline Score).
Time Frame: Baseline and Month 12
Measure: Mean (Standard Error); unit: Resonance raman units (RRU)
Arm/Group | Early Genetic Results Disclosure | Late Genetic Results Disclosure
Number analyzed (Participants) | 56 | 20
Resonance raman units (RRU) | 30,578.3 (653.6) | 31,678.6 (1,066.5)

3. Secondary Outcome: Change in Ocular Carotenoid Status in Response to Genetic Risk Disclosure as Measured by Macular Pigment Optical Volume
Description: Macular Pigment Optical Volume (MPOV) is a unitless measure of the amount of carotenoids present in the macula. Possible scores range from 0 (no carotenoids detected) to greater than 50,000. Change = (Month 12 Score - Baseline Score).
Time Frame: Baseline and Month 12
Measure: Mean (Standard Error); unit: unitless
Arm/Group | Early Genetic Results Disclosure | Late Genetic Results Disclosure
Number analyzed (Participants) | 56 | 20
unitless | 10,622.6 (173.0) | 10,566.1 (290.0)

4. Secondary Outcome: Change in Serum Carotenoid Status in Response to Genetic Risk Disclosure
Description: Serum carotenoid levels are measured in nanograms per milliliter (ng/mL). Possible scores range from 0 (no carotenoids detected) to greater than 1,000. Change = (Month 12 Score - Baseline Score).
Time Frame: Baseline and Month 12
Measure: Mean (Standard Error); unit: nanograms per milliliter (ng/mL)
Arm/Group | Early Genetic Results Disclosure | Late Genetic Results Disclosure
Number analyzed (Participants) | 56 | 20
nanograms per milliliter (ng/mL)
  Lutein + Zeaxanthin | 238.3 (17.2) | 279.2 (29.9)
  Total Carotenoids | 618.0 (47.6) | 818.7 (82.7)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Early Genetic Results Disclosure | Late Genetic Results Disclosure
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/20
Other Adverse Events (participants affected / at risk) | 18/60 | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early Genetic Results Disclosure (N=60) | Late Genetic Results Disclosure (N=20)
Ehlers-Danlos Syndrome hyper-mobility type (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Splenic lesion (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 2 (2) | 1 (1)
Influenza A (Infections and infestations) | 1 (1) | 0 (0)
Elevated cholesterol (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0)
Gout (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Ptosis (Eye disorders) | 1 (1) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Neoplasms benign, malignant and unspecified (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Retinal hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Pruritic rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Our study population was mainly Caucasian because the genetic testing had been validated in this population. Due to logistical constraints, we could not undertake expanded measures of lifestyle modification and coaching, potential active nutritional interventions, or follow-up with individuals in the deferred disclosure group to determine any psychological impact.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-11): https://cdn.clinicaltrials.gov/large-docs/24/NCT05265624/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT05265624/ICF_001.pdf